CLINICAL TRIAL: NCT01059812
Title: A Pan Asian Trial Comparing Efficacy and Safety of NN5401 and Biphasic Insulin Aspart 30 in Type 2 Diabetes (BOOST™: INTENSIFY ALL)
Brief Title: A Pan Asian Trial Comparing Efficacy and Safety of NN5401 and Biphasic Insulin Aspart 30 in Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3597; U1111-1111-7210 (Other: WHO); 101040 (Registry Identifier: JAPIC)
Record Dates: First submitted 2010-01-29; First posted 2010-02-01 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 BID (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected subcutaneously twice daily. Dose was individually adjusted.
  Arms: IDegAsp BID
Drug: biphasic insulin aspart 30 — Injected subcutaneously twice daily. Dose was individually adjusted.
  Arms: BIAsp 30 BID

SUMMARY:
This trial is conducted in Asia. The aim of this clinical trial is to compare NN5401 (insulin degludec/insulin aspart (IDegAsp)) with biphasic insulin aspart (BIAsp) 30 in patients with type 2 diabetes not optimally controlled on once or twice daily insulin with or without metformin.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age (at least 20 years for Japan)
* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Subject on basal human or analogue insulin, once daily (OD) or twice daily (BID) with or without metformin for at least 3 months or subject on premixed human or analogue insulin or self-mixed insulin regimen, containing 20-40% fast/rapid-acting component, OD or BID, with or without metformin, for at least 3 months
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body mass index (BMI) maximum 35.0 kg/m^2

Exclusion Criteria:

* Treatment with oral antidiabetic drugs (OADs) (except metformin) within the last 8 weeks prior to Visit 1
* Treatment with thiazolidinediones (TZDs) or glucagon like peptide 1 (GLP-1) receptor agonists within 3 months prior to Visit 1
* Cardiovascular disease, within the last 6 months prior to Visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer (except basal cell skin cancer or squamous cell skin cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2010-02-01 (Actual); Primary Completion 2010-12-23 (Actual); Study Completion 2010-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (39):
- Novo Nordisk Investigational Site, Shatin, New Territories, Hong Kong
- Japan (15):
  - Novo Nordisk Investigational Site, Chūōku
  - Novo Nordisk Investigational Site, Imizu-shi
  - Novo Nordisk Investigational Site, Kamakura-shi
  - Novo Nordisk Investigational Site, Kashiwara-shi, Osaka
  - Novo Nordisk Investigational Site, Koriyama-shi, Fukushima
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Matsumoto-shi
  - Novo Nordisk Investigational Site, Naha
  - Novo Nordisk Investigational Site, Naka-shi, Ibaraki
  - Novo Nordisk Investigational Site, Oyama-shi, Tochigi
  - Novo Nordisk Investigational Site, Ōita
  - Novo Nordisk Investigational Site, Sapporo-shi, Hokkaido
  - Novo Nordisk Investigational Site, Takatsuki-shi, Osaka
  - Novo Nordisk Investigational Site, Urasoe-shi,
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa
- Malaysia (8):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Georgetown, Penang
  - Novo Nordisk Investigational Site, Johor Bahru
  - Novo Nordisk Investigational Site, Klang, Selangor
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Kota Kinabalu
  - Novo Nordisk Investigational Site, Putrajaya
  - Novo Nordisk Investigational Site, Seremban
- South Korea (11):
  - Novo Nordisk Investigational Site, Ansan
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Guri-si
  - Novo Nordisk Investigational Site, Gyeonggi-do
  - Novo Nordisk Investigational Site, Incheon
  - Novo Nordisk Investigational Site, Jeollanamdo
  - Novo Nordisk Investigational Site, Pusan
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Suwon
  - Novo Nordisk Investigational Site, Wŏnju
- Taiwan (4):
  - Novo Nordisk Investigational Site, Kaohsiung City
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taipei

REFERENCES:
- [Result] Evans M, Gundgaard J, Hansen BB. Cost-Effectiveness of Insulin Degludec/Insulin Aspart Versus Biphasic Insulin Aspart in Patients with Type 2 Diabetes from a Danish Health-Care Perspective. Diabetes Ther. 2016 Dec;7(4):809-823. doi: 10.1007/s13300-016-0195-6. Epub 2016 Aug 23. PMID 27553066
- [Result] Christiansen JS, Niskanen L, Rasmussen S, Johansen T, Fulcher G. Lower rates of hypoglycemia during maintenance treatment with insulin degludec/insulin aspart versus biphasic insulin aspart 30: a combined analysis of two Phase 3a studies in type 2 diabetes. J Diabetes. 2016 Sep;8(5):720-8. doi: 10.1111/1753-0407.12355. Epub 2016 Mar 6. PMID 26612062
- [Result] Taneda S, Hyllested-Winge J, Gall MA, Kaneko S, Hirao K. Insulin degludec/insulin aspart versus biphasic insulin aspart 30 twice daily in insulin-experienced Japanese subjects with uncontrolled type 2 diabetes: Subgroup analysis of a Pan-Asian, treat-to-target Phase 3 Trial. J Diabetes. 2017 Mar;9(3):243-247. doi: 10.1111/1753-0407.12407. Epub 2016 Jul 7. PMID 27059529
- [Result] Haluzik M, Fulcher G, Pieber TR, Bardtrum L, Tutkunkardas D, Rodbard HW. The co-formulation of insulin degludec and insulin aspart lowers fasting plasma glucose and rates of confirmed and nocturnal hypoglycaemia, independent of baseline glycated haemoglobin levels, disease duration or body mass index: A pooled meta-analysis of phase III studies in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jul;20(7):1585-1592. doi: 10.1111/dom.13261. Epub 2018 Mar 25. PMID 29451706
- [Result] Fulcher G, Mehta R, Fita EG, Ekelund M, Bain SC. Efficacy and Safety of IDegAsp Versus BIAsp 30, Both Twice Daily, in Elderly Patients with Type 2 Diabetes: Post Hoc Analysis of Two Phase 3 Randomized Controlled BOOST Trials. Diabetes Ther. 2019 Feb;10(1):107-118. doi: 10.1007/s13300-018-0531-0. Epub 2018 Nov 24. PMID 30474818
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- [Derived] Kaneko S, Chow F, Choi DS, Taneda S, Hirao K, Park Y, Andersen TH, Gall MA, Christiansen JS; BOOST: Intensify All Trial Investigators. Insulin degludec/insulin aspart versus biphasic insulin aspart 30 in Asian patients with type 2 diabetes inadequately controlled on basal or pre-/self-mixed insulin: a 26-week, randomised, treat-to-target trial. Diabetes Res Clin Pract. 2015 Jan;107(1):139-47. doi: 10.1016/j.diabres.2014.09.026. Epub 2014 Oct 14. PMID 25498130
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 45 sites in 5 countries: Japan (16 sites), South Korea (16 sites), Hong Kong (1 site), Malaysia (8 sites) and Taiwan (4 sites).
Groups:
- IDegAsp BID: Insulin degludec/insulin aspart (IDegAsp) was given twice daily (BID) with breakfast and evening meal with or without metformin.
- BIAsp 30 BID: Biphasic insulin aspart (BIAsp 30) was given twice daily (BID) with breakfast and evening meal with or without metformin.
Period: Overall Study
Arm/Group | IDegAsp BID | BIAsp 30 BID
Started | 282 | 142
Exposed | 279 (Three subjects withdrew prior to exposure to trial drug) | 141 (One subject withdrew prior to exposure to trial drug)
Completed | 245 | 126
Not Completed | 37 | 16
Not completed — Adverse Event | 9 | 5
Not completed — Lack of Efficacy | 2 | 2
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal Criteria | 9 | 4
Not completed — Unclassified | 14 | 4

BASELINE CHARACTERISTICS:
Population: Baseline characterises are presented for full analysis set (FAS), which included all randomized subjects. In exceptional cases subjects from the FAS were eliminated; 2 subjects in the IDegAsp group were excluded from the FAS because the subjects were randomized in error in spite of being screening failures.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID | BIAsp 30 BID | Total
Number analyzed (Participants) | 280 | 142 | 422
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.1 (10.2) | 61.2 (9.5) | 59.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 129 | 63 | 192
  Male | 151 | 79 | 230
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.4 (0.8) | 8.4 (0.9) | 8.4 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 7.9 (2.5) | 7.9 (2.5) | 7.9 (2.5)
Body weight at randomisation [Mean (Standard Deviation); unit: kg] | 66.1 (11.2) | 66.0 (11.2) | 66.0 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c (Glycosylated Haemoglobin) After 26 Weeks of Treatment
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF).
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 280 | 142
percentage of glycosylated haemoglobin | -1.38 (0.88) | -1.42 (0.97)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG) at Week 26
Description: Mean of SMPG at 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). For 24 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 265 | 133
mmol/L | 7.6 (1.7) | 7.9 (1.8)

3. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 279 | 141
Episodes/100 years of patient exposure | 956 | 952

4. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes are defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes are defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes are defined as occuring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 279 | 141
Episodes/100 years of patient exposure | 111 | 155

5. Secondary Outcome: Change in Body Weight
Description: Change from baseline in body weight after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 279 | 141
kg | 1.1 (2.9) | 1.4 (3.0)

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp BID | BIAsp 30 BID
Serious Adverse Events (participants affected / at risk) | 23/279 | 12/141
Other Adverse Events (participants affected / at risk) | 84/279 | 39/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=279) | BIAsp 30 BID (N=141)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 1 (1) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Drug toxicity (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Diabetic foot (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Carotid artery occlusion (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=279) | BIAsp 30 BID (N=141)
Diabetic retinopathy (Eye disorders) | 19 (19) | 9 (9)
Nasopharyngitis (Infections and infestations) | 51 (58) | 19 (26)
Upper respiratory tract infection (Infections and infestations) | 21 (24) | 12 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.